CLINICAL TRIAL: NCT04358484
Title: Protocol for a Randomized Pilot Study (FIRST STEPS): Implementation of the Incredible Years-ASLD® Program in Spanish Preschoolers With Autism and Premature Children With Communication or Socialization Difficulties
Brief Title: Implementation of Incredible Years for Autism and Language Delay Program in Spain
Acronym: FS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-220-19
Record Dates: First submitted 2020-03-20; First posted 2020-04-24 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder; Language Delay; Prematurity
Keywords: Autism Spectrum Disorder; Language Delay; Prematurity; Incredible Years; Parenting Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Language Development Disorders; Premature Birth

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from three different sites across Spain: HSJD Barcelona, HGUGM Madrid and HMI Málaga. The first site will recruit parents of premature children and the other two sites will recruit parents of children diagnosed with ASD. Participants who meet inclusion criteria and sign the informed consent will complete a pre-intervention assessment. Families will be randomized to the intervention arm or to the treatment as usual (TAU) group, using stratified randomization regarding cognitive level. Those in the intervention arm will attend the IY-ASLD program and those in the TAU group will continue to receive usual care in their healthcare centers. Due to the COVID-19 pandemic the intervention has been postponed and there will be a re-assessment of parental stress and depressive symptoms in both groups just before starting the intervention. After the IY-ASLD is finished, participants in both groups will complete a post-intervention assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants attend The Incredible Years - ASLD parenting intervention and continue to receive usual care at their healthcare center
  Interventions: Behavioral: Incredible Years - ASD and Language Delay®
- Treatment As Usual (TAU) Group (No Intervention): Participants continue to receive usual care at their Healthcare Center

INTERVENTIONS:
Behavioral: Incredible Years - ASD and Language Delay® — The IY - ASLD Program will consist of 22 weekly online group sessions for parents of children between 2-5 years of age with symptoms or a diagnosis of ASD or delayed language acquisition. The program will be conducted by a therapist and a co-therapist, trained in the model.
  Fidelity to the intervention will be assessed in accordance with the regulations of the program. All of the therapists and co-therapists will be trained in the intervention by accredited trainers. The three main therapists will be supervised by accredited supervisors of the IY Program, seeking accreditation in the intervention. As the intervention IY - ASLD has not been translated into Spanish, the English materials will be used with simultaneous translation into Spanish language.
  Arms: Intervention Group

SUMMARY:
Children with autism spectrum disorders (ASD) usually present coexisting problems in emotion and behavior regulation, similarly as premature children with communication or socialization difficulties. Caring for children with neurodevelopmental difficulties is an important stressor for parents. Therefore, it is essential that families are offered evidence-based interventions at an early stage within the public health service. Group therapy is a cost-effective intervention that can help parents of children diagnosed with autism and those born prematurely. The Incredible Years - ASLD program is an example of this sort of therapy, consisting of a group intervention for parents of preschool children with a diagnosis of ASD or Language Delay. In Spain, group interventions for children with ASD and preterm children presenting with Language Delay are scarce in the public health service. The Incredible Years - ASLD program has not been translated into Spanish and it has not been previously implemented in our country.

The Incredible Years - ASLD group intervention will be carried out in three public Healthcare centers. It is intended to recruit 72 patients diagnosed with ASD or premature children with communication or socialization difficulties, which will be randomized to an Intervention Group or to Treatment as Usual (TAU) Group. The Intervention Group will receive fourteen sessions of the Incredible Years - ASLD program in addition to Treatment as Usual (TAU). In terms of clinical implications, this randomized pilot study could demonstrate the feasibility of implementing this intervention in the regular clinical settings within the Spanish public health service and could be a first step for future controlled studies that demonstrate its effectiveness.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder involving social communication disturbances and a restricted pattern of interests, present before age 3. Premature infants are at particular risk for neurodevelopmental disturbances, such as language delay, difficulties in social communication and ASD.

ASD is often associated with behavior difficulties, emotion regulation difficulties, psychiatric comorbidities and a dysfunctional response to sensory stimuli. Children with premature birth also present difficulties related to emotion and behavior regulation.

Due to these difficulties, caring for children with neurodevelopmental disorders can be very stressful for parents, which could in turn lead to lower effectiveness of interventions and greater mental health difficulties in parents.

Therefore, parenting interventions should not only address children's difficulties, these interventions should also aim to provide support for parents. Since no interventions have specifically addressed these two aspects in the treatment of neurodevelopmental disorders, several therapies have been adapted for this population. This is the case of the intervention at hand: Incredible Years - ASD and Language Delay (IY-ASLD).

In this intervention, in addition to learning strategies to promote the development of skills in children, parents receive support from other parents and from the therapists. The effectiveness of the Incredible Years program has been widely demonstrated in multiple randomized clinical trials, showing an improvement in terms of parental stress levels, depression and parental coping, as well as in children behavior difficulties. Incredible Years is also considered an evidence-based intervention according to the NICE guidelines.

The Incredible Years Program has been adapted for parents of children between ages 2 and 5 diagnosed with ASD, presenting ASD symptoms or language delay. A pilot study conducted in the UK has demonstrated high levels of acceptability, as well as a decrease in levels of parental stress associated with the care of their children. The results of a pilot randomized clinical trial in Wales have been recently published, supporting the feasibility of this intervention in the NHS and showing good levels of acceptability and fidelity to the program and compliance. The Incredible Years - ASLD Program has not been implemented in Spain and to the best of our knowledge it has not been used with parents of children of premature birth with communication and socialization difficulties.

This study aims to demonstrate the feasibility of reliably implementing the IY-ASLD parental program in different outpatient services of the Spanish public health service, as well as exploring its effectiveness in terms of reducing parental distress and improving children outcomes.

The IY - ASLD program will be implemented in three sites across Spain: Hospital Sant Joan de Déu Barcelona (HSJD), Hospital General Universitario Gregorio Marañón (HGUGM) and Hospital Materno Infantil (HMI) de Málaga. In the first site the program will be implemented with parents of premature children with communication and socialization impairment, and in the other two sites the program will be applied with parents of children diagnosed with ASD. The IY-ASLD program will consist of 22 weekly online group sessions for parents of children between 2-5 years of age. The sessions will be conducted by a therapist and a co-therapist, both trained in the program. A total of n = 72 parents (48 with ASD children and 24 with premature children) will be recruited and will be randomized to a control group (36 parents: 24 with ASD children and 12 with premature children) or group intervention (36 parents: 24 with ASD children and 12 with premature children).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria in HGUGM Madrid and HMI Málaga sites:

* Parents who have signed the Informed Consent.
* Parents of children diagnosed with ASD.
* Parents of children between the ages of 2 and 5 years, 11months.
* Fluency in Spanish.

Inclusion criteria in the HSJD Barcelona site:

* Parents who have signed the informed consent.
* Parents of children born with gestational age less than 37 weeks.
* Parents of children with communication or socialization difficulties (Vineland-III scores 1SD below the mean in any of the communication or socialization subdomains).
* Parents of children between the ages of 2 and 5 years, 11months.
* Fluency in Spanish

Exclusion Criteria:

* Attending another structured/manualized parenting program (focused on improving strategies for parents to help their children with behavioral and emotion regulation) at the time of the study.
* Parents of looked after children.

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Autism Program Parent Final Satisfaction Questionnaire | Administered to the intervention group at treatment completion (approximately 22 weeks after baseline).
  Questionnaire for parents assessing their satisfaction with the IY-ASLD Program received.
Register sheet of attendance | Administered to the intervention group weekly throughout treatment (22 weeks total)
  Register of weekly attendance, aimed to determine levels of compliance with the intervention.
Autism Program Parent Weekly Evaluation. | Administered to the intervention group weekly throughout treatment (22 weeks total)
  Questionnaire assessing levels of satisfaction with each therapy session.This survey was specifically developed for the Incredible Years Program and can be found in the Incredible Years manual
Incredible Years® Parent Strategies Questionnaire for Children with Autism (2-5 years) | Administered to the intervention group. Baseline (prior to programme initiation) and immediately after the intervention.
  Questionnaire assessing type of parental strategies specifically aimed at helping children with ASD.

SECONDARY OUTCOMES:
Parental Stress Index (PSI-SF) by Abidin. | Administered to both arms.First assessment before the groups randomization, pre-intervention assessment just before the programme initiation (due to the delay of the intervention because the COVID-19 pandemic), and immediately after the intervention.
  Inventory assessing levels of parental stress regarding the care of their children.
Beck Depression Inventory (BDI) | Administered to both arms. First assessment before the groups randomization, pre-intervention assessment just before the programme initiation (due to the delay of the intervention because the COVID-19 pandemic), and immediately after the intervention.
  Inventory of depressive symptoms for adults, reported by parents.
Autism Specify Five Minutes Speech Sample - ASFMSS | Administered to both arms. Baseline (prior to programme initiation) and immediately after the intervention.
  It measures the construct Expressed emotion in parents of children with neurodevelopmental difficulties.
Alabama Parenting Questionnaire Preschool revision (APQ-Pr). | Administered to both arms. Baseline (prior to programme initiation) and immediately after the intervention.
  It assesses parenting practices, including positive, inconsistent and punitive parenting styles.

OTHER OUTCOMES:
Child Behavior Checklist (CBCL11/2-5), Achenbach. | Administered to both arms. Baseline (prior to programme initiation) and immediately after the intervention.
  List of externalizing, internalizing and total problems. Version for parents of children from 1.5 to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Laia Villalta, Medicine, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Fundació Sant Joan de Déu, Esplugues de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valencia F, Urbiola E, Romero-Gonzalez M, Navas I, Elias M, Garriz A, Ramirez A, Villalta L. Protocol for a randomized pilot study (FIRST STEPS): implementation of the Incredible Years-ASLD(R) program in Spanish children with autism and preterm children with communication and/or socialization difficulties. Trials. 2021 Apr 20;22(1):291. doi: 10.1186/s13063-021-05229-1. PMID 33879224